CLINICAL TRIAL: NCT06122480
Title: Surgical Resection of Synchronous Pulmonary or Hepatic Oligometastatic Pancreatic Ductal Adenocarcinoma (PHOLIPANC): A Phase II Single Arm Trial
Brief Title: Surgical Resection of Synchronous Pulmonary or Hepatic Oligometastatic Pancreatic Ductal Adenocarcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J23143; IRB00414679 (Other: JHM IRB)
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Oligometastatic Disease
Keywords: Hepatic metastasis; Pulmonary metastasis; Oligometastasis; Surgical Resection
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm liver/lung oligometastasis (Experimental): Eligible patients with hepatic or pulmonary oligometastatic adenocarcinoma of the pancreas must have received neoadjuvant FOLFIRINOX chemotherapy in cycles of 14 days, or other clinically indicated alternative. FOLFIRINOX is not a study treatment. Patients with pulmonary metastasis with tumor response or stable disease and a resectable primary tumor after the first 4 cycles can undergo resection of the primary tumor followed by resection of pulmonary metastases or vice versa, if feasible.Patients with hepatic metastasis with tumor response or stable disease and a resectable primary tumor can undergo explorative laparotomy and synchronous resection of the tumor and hepatic metastases, if feasible. In patients who undergo exploratory laparotomy and are deemed to have unresectable disease by the surgeon, the patient may receive 4 more cycles of neoadjuvant chemotherapy 2-4 week after surgery, before the patient will be re-evaluated for the eligibility for the Study Entry Screening.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — All eligible patients with hepatic metastasis will undergo exploratory laparotomy surgery and synchronous resection of the tumor and hepatic metastases, if feasible according to the surgeon, 2-6 weeks after the last neoadjuvant chemotherapy treatment. All eligible patients with pulmonary metastasis will undergo resection of the primary tumor followed by resection of pulmonary metastases or vice versa, if feasible

SUMMARY:
Surgical Resection of Synchronous Pulmonary or Hepatic Oligometastatic Pancreatic Ductal Adenocarcinoma (PHOLIPANC). This is an interventional, open-label, non-randomised, single-arm phase II clinical trial.

Eligible patients with hepatic or pulmonary oligometastatic adenocarcinoma of the pancreas must have received neoadjuvant FOLFIRINOX chemotherapy in cycles of 14 days, or other clinically indicated alternative. FOLFIRINOX is not a study treatment.

DETAILED DESCRIPTION:
In this clinical trial the investigators will enroll subjects with hepatic or pulmonary oligometastatic pancreatic ductal adenocarcinoma and perform a synchronous surgical resection. In patients with progressive disease during or after the first four cycles of neoadjuvant chemotherapy, those patients will not be eligible for study enrollment. Patients with tumor response or stable disease after the first 4-cycles but a non-resectable primary tumor according to the evaluation of an interdisciplinary tumor board must receive 4 more cycles of neoadjuvant chemotherapy before being evaluated for eligibility for the Study Entry Screening. Patients with hepatic metastasis with tumor response or stable disease and a resectable primary tumor after the first 4 cycles can undergo explorative laparotomy and synchronous resection of the tumor and hepatic metastases, if feasible. In patients who undergo exploratory laparotomy and are deemed to have unresectable disease by the surgeon, the patients may receive 4 more cycles of neoadjuvant chemotherapy 2-4 week after surgery, before the patient will be re-evaluated for the eligibility for the Study Entry Screening. Patients with pulmonary metastasis with tumor response or stable disease and a resectable primary tumor after the first 4 cycles can undergo resection of the primary tumor followed by resection of pulmonary metastases or vice versa, if feasible.

All eligible patients with hepatic metastasis will undergo exploratory laparotomy surgery and synchronous resection of the tumor and hepatic metastases, if feasible according to the surgeon, 2-6 weeks after the last neoadjuvant chemotherapy treatment. All eligible patients with pulmonary metastasis will undergo resection of the primary tumor followed by resection of pulmonary metastases or vice versa, if feasible.

ELIGIBILITY:
1. Inclusion Criteria at the Pre-Screening Enrollment

   * Histologically confirmed diagnosis of treatment-naïve limited hepatic or pulmonary metastatic adenocarcinoma of the pancreas Meet the definition of limited hepatic or pulmonary metastasis according to CT/MRI that is done prior to the starting of any anticancer treatment. Either CT scan of chest, abdomen, and pelvis with intravenous contrast or a combination of MRI of abdomen and pelvis and CT scan of chest is acceptable radiographic imaging. CT/MRI can be done at an outside facility, but must be reviewed by a Johns Hopkins Medicine radiologist.
   * Measurable disease according to RECIST v1.1
   * Eastern Cooperative Oncology Group (ECOG) performance status 0-1
   * Being a candidate for the chemotherapy with FOLFIRINOX or modified FOLFIRINOX
   * Patients ≥18 years at the time of signing the informed consent
   * Patient's written informed consent prior to any trial-specific procedure
   * Patient's legal capacity to consent to participation in the clinical trial
2. Exclusion Criteria at the Pre-Screening Enrollment

   * Acinar cell carcinoma and/or neuroendocrine carcinoma of the pancreas
   * Symptomatic clinically significant ascites
   * Evidence of any distant metastases other than limited hepatic or pulmonary metastasis as defined in inclusion criterion 1.
   * Evidence of simultaneous pulmonary and hepatic metastases
   * Any tumor-specific pretreatment of the adenocarcinoma of the pancreas (including but not limited to surgery, radiation therapy, chemotherapy or ablative procedures). Currently being on FOLFIRINOX or modified FOLFIRINOX (mFOLFIRINOX) is allowed, unless more than 2 treatments of FOLFIRINOX or mFOLFIRINOX has been given.
   * Any malignancies other than adenocarcinoma of the pancreas in the 2 years before the start of the clinical trial except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, breast cancer, prostate cancer or superficial bladder tumors (Ta, Tis and T1)
   * Known HIV seropositivity
   * Known active or chronic Hepatitis B or Hepatitis C infection
   * Any other severe concomitant disease or disorder, which could influence patient's ability to participate in the clinical trial and his/her safety during the trial or interfere with interpretation of results, e.g., severe hepatic, renal, pulmonary, cardiovascular, metabolic or psychiatric disorders

3.2 Eligibility Criteria for Study Entry Enrollment at the Pre-Surgery phase 3.2.1 Inclusion Criteria for study continuation at the Pre-Surgery phase

* ECOG performance status 0-1
* Received FOLFIRINOX, modified FOLFIRINOX or the further modified forms including FOLFIRI, FOLFOX, 5FU or capecitabine. Liposomal irinotecan is permitted. Switching to gemcitabine/nal-paclitaxel due to intolerability of FOLFIRINOX is also permitted.
* Radiographical evidence of disease response or stable disease with CA19-9 decrease > 20% from the baseline or CA19-9 that is not detectable
* Patients ≥18 years at the time of signing the informed consent
* Patient's written informed consent prior to any trial-specific procedure
* Patient's legal capacity to consent to participation in the clinical trial

3.2.2 Exclusion Criteria for Study Entry Enrollment at the Pre-surgery phase

* Symptomatic clinically significant ascites
* Evidence of any distant metastases other than limited hepatic or pulmonary metastasis as defined in inclusion criterion 1.
* Evidence of simultaneous pulmonary and hepatic metastases
* Any malignancies other than adenocarcinoma of the pancreas in the 2 years before the start of the clinical trial except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, breast cancer, prostate cancer or superficial bladder tumors (Ta, Tis and T1)
* Pregnant or breast-feeding female
* Radiographic evidence of severe portal hypertension
* Liver cirrhosis ≥ Child Pugh B
* Known HIV seropositivity
* Active or chronic Hepatitis B or Hepatitis C infection
* Clinically significant cardiovascular or vascular disease or disorder ≤6 months before enrolment into the clinical trial (e.g., myocardial infarction, unstable angina pectoris, chronic heart failure New York Heart Association (NYHA) ≥ Grade 2, uncontrolled arrhythmia, cerebral infarction)
* Any other severe concomitant disease or disorder, which could influence patient's ability to participate in the clinical trial and his/her safety during the trial or interfere with interpretation of results, e.g., severe hepatic, renal, pulmonary, cardiovascular, metabolic or psychiatric disorders.
* Hepatic metastasis that are only amenable to ablation. However, if liver lesions are found intraoperatively and subsequently ablated and if the pancreatic surgery is distal pancreatectomy, the patients would still be considered evaluable. Ablation of liver lesions during the pancreatoduodenectomy is not allowed.
* Radiographical evidence of disease progression.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
2-year overall survival will be measured for the evaluable liver and Lung oligometastasis patient cohorts, respectively, and compare to historical controls. | 48 months
  Time-to-event data will be analyzed according to the Kaplan-Meier method (product-limit analysis). Patients who are not known to have had an event by the time of the analyses will be censored based on the last recorded date the patient was known to be event-free.
Compare the Intrametastasis effector T cell infiltration | 48 months
  The liver oligometastasis cohort and the lung oligometastasis cohort will be compared in terms of intra-tumoral CD8+ T cells.

SECONDARY OUTCOMES:
Perioperative morbidity and mortality as assessed by the Common terminology criteria for adverse events | 48 months
  The safety analysis includes type, incidence, and severity of adverse events (severity according to Common terminology criteria for adverse events version 5.0).
Medium Overall Survival (OS) and Disease Free Survival | 48 months
  Kaplan-Meier survival curves will be constructed to summarize disease free survival and overall survival, respectively.
Health-related quality of life will be assessed by the European organization for research and treatment of cancer quality of life questionnaire (EORTC QLQ-C30) | 48 months
  Questions 1 to 28, a 4-point scale is used, ranging from 1 ("Not at all") to 4 ("Very much"), with lower scores indicating a more positive outcome. Questions 29 and 30 employ a 7-point scale, with scores ranging from 1 ("Very poor") to 7 ("Excellent"), where higher scores signify a better outcome
Health-related quality of life as assessed by the European Organisation for Research and Treatment of Cancer in Pancreatic Cancer (EORTC QLQ-PAN26) | 48 months
  European Organisation for Research and Treatment of Cancer in pancreatic cancer includes 26 questions with two subscales: functioning scales (4 questions),and symptom scales (22 questions). The functional scale, the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life. All scores are scaled to range from 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Jin He, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No